CLINICAL TRIAL: NCT00966030
Title: An Open-Label, Randomized, 2-Period Crossover Study to Demonstrate the Definitive Bioequivalence of a Single Dose of a Tablet Form of MK0974 Ethanolate Vs. a Single Dose of the Reference MK0974 Liquid Filled Capsule in Healthy Subjects
Brief Title: Bioequivalence of the Tablet and Liquid-Filled Capsule Forms of MK0974 (0974-042)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0974-042; MK0974-042; 2009_649
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MK0974 Tablet
  Interventions: Drug: MK0974 tablet
- 2 (Active Comparator): MK0974 Liquid filled capsule
  Interventions: Drug: Comparator: MK0974 liquid filled capsule

INTERVENTIONS:
Drug: MK0974 tablet — MK0974 280 mg tablet in one of two treatment periods
  Arms: 1
Drug: Comparator: MK0974 liquid filled capsule — MK0974 300 mg liquid filled capsule in one of two treatment periods
  Arms: 2

SUMMARY:
This study will demonstrate the definitive bioequivalence of a solid dose formulation of MK0974 to the liquid filled capsule formulation of MK0974.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a nonsmoker
* Subject is willing to comply with the study restrictions

Exclusion Criteria:

* Subject has history of stroke, chronic seizures, or any major neurological disorder
* Subject has a history of cancer
* Subject is a nursing mother
* Subject has uncontrolled high blood pressure
* Subject has or has a history of any disease or condition that might made participation in the study unsafe or confound the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC(0 to infinity)) following single dose administration of MK0974 tablet formulation and MK0974 liquid filled capsule formulation | Through 48 Hours Post Dose
Peak plasma concentration (Cmax) following single dose administration of MK0974 tablet formulation and MK0974 liquid filled capsule formulation | Through 48 Hours Post Dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC